CLINICAL TRIAL: NCT04721093
Title: Effects and Safety Evaluation of Changes in Cognitive Function of Photobiomodulation Treatment for Patients With Mild Cognitive Impairment (MCI): Single-institutional Prospective Clinical Trial, Single Group, Pilot Trial
Brief Title: Effects of Photobiomodulation on Changes in Cognitive Function and rCBF in MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Head of Rehabilitation Medicine, Principal Investigator, Pusan National University Yangsan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-2018-006
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Regional Cerebral Blood Flow; Mild Cognitive Impairment; Cognitive Function
Keywords: Photobiomodulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Patients with Mild Cognitive Impairment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PBM(Photobiomodulation) (Experimental): Subjects applied PBM(Color-DNA-WSF U, Color Seven; 610 nm±10nm wavelength; 3.0 mW/㎠±20%) therapy in the locations of the sternocleidomastoid muscle in the ICA area and the trapezius muscle in VA area. PBM was applied 5 times a week for 8 weeks, 30 minutes per session.
  Interventions: Device: Photobiomodulation device

INTERVENTIONS:
Device: Photobiomodulation device — In this study, PBM was applied using a machine made to be attached to the subject in the form of a probe. In this clinical trial, a low-intensity irradiation device (Color-DNA-WSF U) from Color seven was used to deliver visible light (610nm± 10nm wavelength, 3.0mW/㎠±20%) irradiation. PBM was applied 5 times a week for 8 weeks, 30 minutes per session.
  Other Names: Low level light theraphy

SUMMARY:
This pilot study has two goals. The first is to see if the cognitive improves when VA and CA are stimulated in MCI patients, and the second is to do an explanatory data analysis to see if that improves cognitive in relation to the rCBF improvement.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed codsent sill undergo a 1 day screening period to determine eligibility for study entry. Subjects who pass the screening test will receive a registration number within 7 days and proceed with the pre-intervention test as follows.

ELIGIBILITY:
Inclusion Criteria:

* The patients with mild cognitive impairment(MCI). The MCI was diagnosed based on medical history and neurological examination
* A sufficient level of education to understand study procedures and be able to communicate with site personnel

Exclusion Criteria:

* Any psychiatric disorders such as schizophrenia that would compromise participation
* Those with central nervous system disease
* Serious cognitive problems(MoCA score 7 or less).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Korean Version of Montreal Cognitive Assessment(MoCA) score change | Baseline and week 8
  The MoCA is a validated, instrument assessing overall cognitive function in patients with mild cognitive impairment. Possible scores range from 0 to 30(Higher numbers indicate better cognitive function). Change=(week 8 score-baseline score).
Single photon emission computed tomography(SPECT) z-score change | Baseline and week 8
  The SPECT is a validated, instrument assessing regional Cerebral Blood Flow(rCBF). Possible scores range from -6.5 to 6.5. The score indicates how far the data value is from the means for each region from the normal database. Change=(week 8 score-baseline score).
The verbal learning test(VLT) score change | Baseline and week 8
  The VLT is a validated, instrument assessing memory domain. The VLT is a task in which the examiner reads 12 words and the subject is immediately asked to remember as many words as possible. Possible scores range from 0 to 12(Higher numbers indicate better). Change=(week 8 score-baseline score).
The trail making test(TMT) score change | Baseline and week 8
  The TMT is a validated, instrument assessing frontal/executive functions domain, requires the subject to draw a line that alternates between numbers and days of the week in a consecutive manner.
  The score is calculated by subtracting the number of errors from the total time it took to complete the test. And the score is converted to %ile(0 to 100) based on the normal database and changed(Higher numbers indicate better). Change=(week 8 score-baseline score).
Boston naming test(BNT) score change | Baseline and week 8
  The BNT is a validated, instrument assessing visual confrontation naming. BNT assesses the naming ability using 60 black and white images that are organized. The subject is asked to name what is depicted in the image. Possible scores range from 0 to 60(Higher numbers indicate better). Change=(week 8 score-baseline score).
Rey complex figure test(RCFT)-'copy' score change | Baseline and week 8
  The RCFT 'copy' is a validated, instrument assessing visuo-constructive abilities. The RCFT 'copy' requires the subject to observe and replicate an image. The score is scored as 0, 0.5, 1 or 2 for each of the 18 factors. Point 2 is when the shape and position of the element is accurately drawn, point 1 is when one of the shape or position is correct. Point 0.5 is when both the shape and position are incorrect, but the examinee can determine what the subject was trying to draw, and point 0 is the case when the shape and position difference are both inadequate, and when the element is not drawn. The total score is the sum of the scores scored for each of the 18 elements; It is possible scores range from 0 to 36(Higher numbers indicate better). Change=(week 8 score-baseline score).
Rey complex figure test(RCFT)-'Immediate Recall' score change | Baseline and week 8
  The RCFT 'immediate recall' is a validated, instrument assessing visuo-constructive memory abilities. The RCFT 'immediate recall' requires the subject to flip the page and replicate the image. The score is scored as 0, 0.5, 1 or 2 for each of the 18 factors. Point 2 is when the shape and position of the element is accurately drawn, point 1 is when one of the shape or position is correct. Point 0.5 is when both the shape and position are incorrect, but the examinee can determine what the subject was trying to draw, and point 0 is the case when the shape and position difference are both inadequate, and when the element is not drawn. The total score is the sum of the scores scored for each of the 18 elements; It is possible scores range from 0 to 36(Higher numbers indicate better). Change=(week 8 score-baseline score).

CONTACTS AND LOCATIONS:
Overall Officials: Yong-il Shin, PhD, Study Director — Pusan National University Yangsan Hospital
Locations (1):
- Pusan national university Yangsan Hospital, Gyeongsang, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No